CLINICAL TRIAL: NCT01944969
Title: Interventional, Open-label, Long-term Extension Study to Evaluate the Safety and Tolerability of Brexpiprazole as Adjunctive Treatment in Patients With Major Depressive Disorder
Brief Title: Long-term Safety and Tolerability Study of Brexpiprazole as Adjunctive Treatment in Patients With Major Depressive Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because the lead-in study (14571A) in elderly was terminated; see Detailed Description.
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14767B; 2012-004169-42 (EudraCT Number)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 1, 2, or 3 mg/day, once daily dose, tablets, orally. Uptitration in weekly steps from 0.5 mg/day (patients ≥65) or 1 mg/day (patients 18-64 years)

SUMMARY:
To evaluate the long-term safety and tolerability of brexpiprazole as adjunctive treatment in patients with Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
This extension safety study was terminated early because one of the lead-in studies (14571A) in elderly was terminated and because the Sponsor considered that sufficient long-term safety data has already been collected in the development programme in the population aged 18-65 yrs.

ELIGIBILITY:
Inclusion Criteria:

* The patient is judged to benefit from adjunctive treatment with brexpiprazole according to the clinical opinion of the investigator.
* The patient had MDD at entry in lead-in brexpiprazole studies, NCT01838681 / 14570A or NCT01837797 / 14571A, diagnosed according to DSM-IV-TR™.
* The patient agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* The patient has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The patient has been diagnosed with a psychiatric disorder other than MDD during the lead-in studies NCT01838681 / 14570A or NCT01837797 / 14571A.
* The patient, in the opinion of the investigator or according to C-SSRS, is at significant risk of suicide.
* The patient has any relevant medical history or current presence of systemic disease.
* The patient has, at the Baseline Visit an abnormal ECG that is, in the investigator's opinion, clinically significant.
* The patient has a moderate or severe ongoing adverse event related to study medication from the lead-in studies considered of potential safety risk by the investigator.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- US008, Orlando, Florida, United States

REFERENCES:
- See also: EudraCT (EMA) Result Posting — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-004169-42/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Brexpiprazole and ADT: Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Brexpiprazole: 1, 2, or 3 mg/day, once daily dose, tablets, orally
Period: Overall Study
Arm/Group | Brexpiprazole and ADT
Started | 26
Completed | 0
Not Completed | 26
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Non-compliance with IMP | 1
Not completed — Administrative or other reasons | 23

BASELINE CHARACTERISTICS:
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.12 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 14
  Slovakia | 2
  Sweden | 2
  United Kingdom | 1
  Estonia | 3
  Finland | 2
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of participants with Treatment-Emergent Adverse Events
Time Frame: From baseline to Week 52
Measure: Number; unit: participants
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 26
participants | 28

2. Primary Outcome: Number of Withdrawals
Description: Number of withdrawals
Time Frame: From baseline to Week 52
Population: 26 patients were withdrawn; the reason for withdrawal was not poor tolerability, but mainly (23 patients) because the study was terminated. Please see withdrawn reasons in the participant flow section for the other reasons.
Measure: Number; unit: participants
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 26
participants | 26

3. Secondary Outcome: Number of Patients With Risk of Suicidality Assessed Using the Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
Description: The Columbia Suicide Severity Rating Scale (eC-SSRS) is a semi-structured interview developed to systematically assess suicidal ideation and behaviour of patients participating in a clinical study. The C-SSRS has 5 questions addressing suicidal ideation, 5 sub-questions assessing the intensity of ideation, and 4 questions addressing suicidal behaviour. The electronic C-SSRS (eC-SSRS) is a patient-rated electronic version using interactive voice response technology. A structured CSSRS script of standardised questions, follow-up prompts, error-handling and scoring conventions is used for administration.
Time Frame: From baseline to Week 52
Population: all-patients treated set (APTS)
Measure: Number; unit: participants
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 26
participants
  No suicidal ideation or behaviour | 25
  Any non-suicidal self-injurious behavior | 0
  Suicidal Ideation | 1
  Preparatory action towards imminent suicidal | 0
  Not fatal suicide attempt | 0
  Completed suicide | 0

4. Secondary Outcome: Change in Depressive Symptoms
Description: The Montgomery and Aasberg Depression Rating Scale (MADRS) total score
Time Frame: From baseline to Week 52
Population: None of the patients completed the study. A total of 26 patients were enrolled when the study was prematurely terminated(Planned: 1184 patients). No data were collected because none of the 26 patients that were enrolled completed the study because of early termination.
Groups:
- Brexpiprazole and ADT: Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Brexpiprazole: 1,2, or 3 mg/day, once daily dose, tablets, orally
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Patients in Remission
Description: Based on a pre-specified MADRS total score
Time Frame: From baseline to Week 52
Population: No patients completed the study. Only 26 patients were enrolled at prematurely study termination (Planned: 1184 patients). No data were collected because none of the 26 patients that were enrolled completed the study because of early termination.
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Clinical Global Impression
Description: Clinical Global Impression - Severity of illness (CGI-S) score
Time Frame: From baseline to Week 52
Population: as for outcome 5
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Health-related Quality of Life
Description: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-(SF)) total score
Time Frame: From baseline to Week 52
Population: as for outcome 5
Arm/Group | Brexpiprazole and ADT
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Health-related Quality of Life
Description: The EuroQoL 5 Dimensions 5L version (EQ-5D-5L) Visual Analogue Scale (VAS) is a patient-reported assessment designed to measure the patient's wellbeing. It consists of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a visual analogue scale (VAS) of the overall health state. Each descriptive item is rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems) and a single summary index (from 0 to 1) can be calculated. The VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and Week 52
Population: as for outcome 5
Groups:
- Brexpiprazole: Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Brexpiprazole: 1, 2, or 3 mg/day, once daily dose, tablets, orally
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From baseline to Week 52
Arm/Group | Brexpiprazole and ADT
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 5/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole and ADT (N=26)
Accidental overdose (Injury, poisoning and procedural complications) | 3
Lethargy (Nervous system disorders) | 2

LIMITATIONS AND CAVEATS:
Because the study was terminated, few efficacy data were collected. These data have not been reported in accordance with the ICH E3 regarding abbreviated clinical study reports. Furthermore, no firm conclusions can be drawn regarding safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No